CLINICAL TRIAL: NCT06051019
Title: Comparison Between the Effects on Fatigue of Aerobic Training Versus Balance Training in Patients With Multiple Sclerosis: a Randomised Crossover Trial.
Brief Title: Effect of Aerobic Training vs Balance Training on Fatigue Symptom in Multiple Sclerosis Patient (FATI-gate)
Acronym: FATI-gate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24C601
Record Dates: First submitted 2023-07-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: fatigue; balance; multiple sclerosis; aerobic training; balance training
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training (FIRST), then balance training (SECOND) (Experimental): Crossover trial: aerobic training (first treatment), then balance training (second treatment).
  Interventions: Other: Aerobic training; Other: Balance training
- Balance training (FIRST), then aerobic training (SECOND) (Experimental): Crossover trial: balance training (first treatment), then aerobic training (second treatment).
  Interventions: Other: Aerobic training; Other: Balance training

INTERVENTIONS:
Other: Aerobic training — Aerobic training: 15 daily sessions (5 sessions per week), each lasting approximately 90 minutes. Sessions will be performed with the assistance or supervision of a physical therapist and will consist of the following steps: 1) warm up with a stationary bike (no load, 10 min, 60 cycles/min); 2) upper and lower limb stretching (10 min); 3) 10 min rest in a sitting position; 4) first exercise bout: stationary bike, 15 min, 60 cycles/min (the load will be modulated so that the participant's heart rate is between 60 and 70% of the estimated maximum heart rate, and the patient perceives moderate fatigue on the Borg Rating of Perceived Exertion; 5) upper and lower limb stretching (10 min); 6) 10 min rest in a sitting position; 7) second exercise bout (same parameters as the first exercise bout); 8) upper and lower limb stretching (10 min).
Other: Balance training — Balance training: 15 daily sessions (5 sessions per week), each lasting approximately 90 minutes. Treatments will be performed with a physical therapist and will consist of the following exercises: 1) standing with feet together, 2) standing with closed eyes, 3) standing on unstable surfaces, 4) standing while performing upper limbs movements; 5) standing while performing head rotations; 6) walking on a treadmill at alternating speeds; 7) leg press and chest press exercises for training trunk balance during ballistic movements of the upper and lower limbs. These constituents of balance training can be combined in the same task according to the participant's ability.

SUMMARY:
Fatigue and impaired balance frequently affect patients with Multiple Sclerosis (MS). This is an open, prospective randomised crossover trial aimed at clarifying whether an improvement in balance control after balance training would also improve fatigue in patients with MS. Balance training will be compared to aerobic training, which is known to be effective on fatigue.

DETAILED DESCRIPTION:
Fatigue is known to affect patients with Multiple Sclerosis (MS), with a prevalence ranging from 55% to 83%, thus contributing to the level of disability, compromising the Quality of Life, and increasing the overall treatment costs. For these reasons, fatigue is considered a main target for pharmacological and non-pharmacological therapies for MS.

The physiopathology of fatigue in MS is still not completely understood, and previous research has shown correlations with reduced motor performance, disease progression and depression. Some possible mechanisms of fatigue in MS have been hypothesised but not yet proven, such as structural alterations in the central nervous system, altered immune function in the brain, impaired pituitary gland function, and changes in cardiac or muscle activity.

Patients with MS also frequently show balance impairments, with prevalence peaking at 87.9%, and previous studies have suggested a causal relationship between fatigue and balance deficits.

Therapeutic exercise has shown a key role in contrasting the functional decline and disability secondary to MS. Several studies have evaluated the effects of different types of training, such as balance training and aerobic training, on balance impairment and the overall patient's functional performance.

In the literature, it is not uncommon to observe improvements in fatigue after the administration of exercise therapy targeted at the balance impairment. However, the literature has not yet clarified whether an improvement in balance control after balance training would also result in an improvement in the scales used to measure fatigue.

The aim of this open prospective randomised crossover trial is to compare the effects of two different types of therapeutic exercise, aerobic training (AT) and balance training (BT), in modifying the intensity of fatigue in patients with MS. AT and BT will be administered at different times to the same patients (crossover trial). Both AT and BT will consist of 15 treatment sessions (5 sessions per week). Patients with MS will be randomly assigned to AT or BT in the first treatment period and then switched to the other type of training in the second treatment period. The time interval between the two time periods will last 60 days, during which the patients will not perform any physical exercise.

In each treatment period, the participants will perform three measurement sessions: before intervention (T0), at the end of intervention (T1), and 30 days after the end of intervention (T2).

ELIGIBILITY:
Inclusion criteria:

* MS diagnosis according to the revised McDonalds criteria. Relapsing-remitting, primary and secondary progressive MS forms are allowed;
* Expanded Disability Status Scale (EDSS) between 2 and 6, included;
* Fatigue as indicated by a total score of mFIS ≥ 20/84;
* Balance impairment as indicated by a performance at the Equitest Sensory Organisation Test below age-matched normal values (95th percentile of control values).

Exclusion criteria:

* Any of the following in the month before enrolment: an MS relapse; current corticosteroids therapy because of MS; change in medicines prescribed against fatigue; attending an intensive physical therapy program;
* New or active lesions on a brain or spinal cord MRI scan in the 12 months before the study enrolment;
* Angioplasty for chronic cerebrospinal venous insufficiency in the six months before enrolment;
* Any musculoskeletal disease or any additional neurological disorder which causes by itself a balance or gait impairment;
* Any other condition causing fatigue by itself;
* Any unstable cardiological disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale Italian version | The Modified Fatigue Impact Scale was assessed: before intervention, at end of first intervention, 30 days after end of first intervention, before second intervention, at end of second intervention, 30 days after end of second intervention
  Modified Fatigue Impact Scale (mFIS) Italian version: The Modified Fatigue Impact Scale is a self-administered questionnaire comprising 21 items assessing how often fatigue interferes with everyday life. Modified Fatigue Impact Scale score ranges from 0 to 84, with higher scores indicating more fatigue.

SECONDARY OUTCOMES:
Equiscale | The Equiscale was assessed: before intervention, at end of first intervention, 30 days after end of first intervention, before second intervention, at end of second intervention, 30 days after end of second intervention
  Equiscale: The Equiscale is an eight-item rating scale developed to measure balance in Multiple Sclerosis. Each item is scored on three categories. Scores range from 0 to 16, with higher scores indicating better balance.
Equitest® Sensory Organization Test | The Sensory Organization Test was computed: before intervention, at end of first intervention, 30 days after end of first intervention, before second intervention, at end of second intervention, 30 days after end of second intervention
  Equitest Sensory Organization Test (SOT): The Equitest Sensory Organization Test is a posturography test, assessing six different balance conditions. From the six balance tasks, a composite score is obtained from the amplitude of the centre of mass sway during standing, ranging from 0 (i.e., falling) to 100 (i.e., perfect stability), with higher scores indicating better balance.
Gait speed | The gait speed was assessed: before intervention, at end of first intervention, 30 days after end of first intervention, before second intervention, at end of second intervention, 30 days after end of second intervention
  Gait speed measured from the 10-meter walking test.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Perucca, MD, Study Chair — Istituto Auxologico Italiano; Antonio Caronni, MD, Principal Investigator — Istituto Auxologico Italiano; Stefano Scarano, MD, Principal Investigator — Istituto Auxologico Italiano; Antonio Robecchi Majnardi, MD, Principal Investigator — Istituto Auxologico Italiano; Giovanna Russo, MD, Principal Investigator — Istituto Auxologico Italiano

REFERENCES:
- [Background] Bakshi R, Shaikh ZA, Miletich RS, Czarnecki D, Dmochowski J, Henschel K, Janardhan V, Dubey N, Kinkel PR. Fatigue in multiple sclerosis and its relationship to depression and neurologic disability. Mult Scler. 2000 Jun;6(3):181-5. doi: 10.1177/135245850000600308. PMID 10871830
- [Background] Brichetto G, Piccardo E, Pedulla L, Battaglia MA, Tacchino A. Tailored balance exercises on people with multiple sclerosis: A pilot randomized, controlled study. Mult Scler. 2015 Jul;21(8):1055-63. doi: 10.1177/1352458514557985. Epub 2014 Nov 12. PMID 25392337
- [Background] Flachenecker P, Kumpfel T, Kallmann B, Gottschalk M, Grauer O, Rieckmann P, Trenkwalder C, Toyka KV. Fatigue in multiple sclerosis: a comparison of different rating scales and correlation to clinical parameters. Mult Scler. 2002 Dec;8(6):523-6. doi: 10.1191/1352458502ms839oa. PMID 12474995
- [Background] Giesser BS. Exercise in the management of persons with multiple sclerosis. Ther Adv Neurol Disord. 2015 May;8(3):123-30. doi: 10.1177/1756285615576663. PMID 25941539
- [Background] Giovannoni G. Multiple sclerosis related fatigue. J Neurol Neurosurg Psychiatry. 2006 Jan;77(1):2-3. doi: 10.1136/jnnp.2005.074948. PMID 16361582
- [Background] Hebert JR, Corboy JR. The association between multiple sclerosis-related fatigue and balance as a function of central sensory integration. Gait Posture. 2013 May;38(1):37-42. doi: 10.1016/j.gaitpost.2012.10.015. Epub 2012 Nov 28. PMID 23200463
- [Background] Hebert JR, Corboy JR, Manago MM, Schenkman M. Effects of vestibular rehabilitation on multiple sclerosis-related fatigue and upright postural control: a randomized controlled trial. Phys Ther. 2011 Aug;91(8):1166-83. doi: 10.2522/ptj.20100399. Epub 2011 Jun 16. PMID 21680771
- [Background] Khan F, Amatya B, Galea M. Management of fatigue in persons with multiple sclerosis. Front Neurol. 2014 Sep 15;5:177. doi: 10.3389/fneur.2014.00177. eCollection 2014. PMID 25309504
- [Background] Kos D, Kerckhofs E, Carrea I, Verza R, Ramos M, Jansa J. Evaluation of the Modified Fatigue Impact Scale in four different European countries. Mult Scler. 2005 Feb;11(1):76-80. doi: 10.1191/1352458505ms1117oa. PMID 15732270
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Larson RD. Psychometric properties of the modified fatigue impact scale. Int J MS Care. 2013 Spring;15(1):15-20. doi: 10.7224/1537-2073.2012-019. PMID 24453758
- [Background] Mayo NE, Bayley M, Duquette P, Lapierre Y, Anderson R, Bartlett S. The role of exercise in modifying outcomes for people with multiple sclerosis: a randomized trial. BMC Neurol. 2013 Jun 28;13:69. doi: 10.1186/1471-2377-13-69. PMID 23809312
- [Background] Mills RJ, Young CA. The relationship between fatigue and other clinical features of multiple sclerosis. Mult Scler. 2011 May;17(5):604-12. doi: 10.1177/1352458510392262. Epub 2010 Dec 6. PMID 21135018
- [Background] Mostert S, Kesselring J. Effects of a short-term exercise training program on aerobic fitness, fatigue, health perception and activity level of subjects with multiple sclerosis. Mult Scler. 2002 Apr;8(2):161-8. doi: 10.1191/1352458502ms779oa. PMID 11990874
- [Background] Rampello A, Franceschini M, Piepoli M, Antenucci R, Lenti G, Olivieri D, Chetta A. Effect of aerobic training on walking capacity and maximal exercise tolerance in patients with multiple sclerosis: a randomized crossover controlled study. Phys Ther. 2007 May;87(5):545-55. doi: 10.2522/ptj.20060085. Epub 2007 Apr 3. PMID 17405806
- [Background] Rota V, Perucca L, Simone A, Tesio L. Walk ratio (step length/cadence) as a summary index of neuromotor control of gait: application to multiple sclerosis. Int J Rehabil Res. 2011 Sep;34(3):265-9. doi: 10.1097/MRR.0b013e328347be02. PMID 21629125
- [Background] Stankoff B, Waubant E, Confavreux C, Edan G, Debouverie M, Rumbach L, Moreau T, Pelletier J, Lubetzki C, Clanet M; French Modafinil Study Group. Modafinil for fatigue in MS: a randomized placebo-controlled double-blind study. Neurology. 2005 Apr 12;64(7):1139-43. doi: 10.1212/01.WNL.0000158272.27070.6A. PMID 15824337
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Background] Tesio L, Perucca L, Franchignoni FP, Battaglia MA. A short measure of balance in multiple sclerosis: validation through Rasch analysis. Funct Neurol. 1997 Sep-Oct;12(5):255-65. PMID 9439943
- [Background] Tesio L, Rota V, Longo S, Grzeda MT. Measuring standing balance in adults: reliability and minimal real difference of 14 instrumental measures. Int J Rehabil Res. 2013 Dec;36(4):362-74. doi: 10.1097/MRR.0000000000000037. PMID 24185405